CLINICAL TRIAL: NCT00205543
Title: Role of Suture Closure in Post-Operative Uvulopalatopharyngoplasty Outcomes
Brief Title: Study of Effects of Sutures on Results of Palate Surgery for Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03802
Record Dates: First submitted 2005-09-15; First posted 2005-09-20 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; airway obstruction; sleep-disordered breathing
MeSH Terms: conditions — Sleep Apnea, Obstructive; Airway Obstruction; Sleep Apnea Syndromes | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): suture palate after resection
  Interventions: Procedure: uvulopalatopharyngoplasty with or without sutures
- 2 (Experimental): suture one side of palate afer resection
  Interventions: Procedure: uvulopalatopharyngoplasty with or without sutures
- 3 (Experimental): no sutures in palate after resection
  Interventions: Procedure: uvulopalatopharyngoplasty with or without sutures

INTERVENTIONS:
Procedure: uvulopalatopharyngoplasty with or without sutures — standard UPPP

SUMMARY:
In this study we will examine whether suture repair of the palate, or roof of mouth, has any effect on results of palate surgery performed for treatment of obstructive sleep apnea.

DETAILED DESCRIPTION:
Uvulopalatopharyngoplasty, or UPPP, is the most common surgical procedure performed for the treatment of obstructive sleep apnea. The procedure involves removal of redundant tissue from the lower palate (roof of mouth), including the uvula, and then suturing the cut edges of the remaining tissue together. However it is frequently noted by surgeons that sutures placed in the roof of the mouth do not stay intact. Also, in standard tonsillectomy, which involves removal of the tonsils and thus creation of a wound near the palate, no suturing is used, which does not seem to affect how the area heals. Previous studies have shown no significant differences in complication rates, post-operative pain, or symptom outcomes in patients undergoing tonsillectomy either with or without suture repair of the tonsillectomy wound. In this study we will examine whether suture repair following UPPP has any effect on post-operative pain, healing, or treatment success in terms of symptom resolution or post-operative sleep study results.

ELIGIBILITY:
Inclusion Criteria:

* sleep-study documented obstructive sleep apnea
* sleep apnea refractory to non-surgical treatments including continuous positive airway pressure (CPAP)
* age > 21

Exclusion Criteria:

* previous palate surgery

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
sleep study result at 3-6 months; symptom changes at 3-6 months; pain at 0-3 weeks; post-operative complications at any time; post-operative anatomic result/appearance at 3-6 months | 6-12mo

SECONDARY OUTCOMES:
Operative time | immediate
Procedure cost | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Evan R Reiter, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Department of Otolaryngology - Head & Neck Surgery, Virginia Commonwealth University, Richmond, Virginia, United States